CLINICAL TRIAL: NCT05364957
Title: Intragastric Balloon in Obese Patients With Uncontrolled Asthma: a Multicentre Randomized Controlled Study
Brief Title: Intragastric Balloon in Obese Patients With Uncontrolled Asthma
Acronym: BOA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/18/0473; 2019-A00595-52 (Other: ANSM)
Record Dates: First submitted 2022-04-21; First posted 2022-05-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Asthma
Keywords: Intra Gastric Balloon; uncontrolled asthma; Obesity with asthma
MeSH Terms: conditions — Obesity; Asthma | interventions — Diet

STUDY DESIGN:
Intervention Model Description: The patients will be randomly assigned either to the group treated with IGB combined with diet and exercise or the group treated with diet and exercise alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (PEC dietary hygiene) (Other): Diet and exercise alone (control)
  Interventions: Procedure: Dietary; Procedure: Exercise intervention
- Experimental (BIG + PEC dietary hygiene) (Experimental): Intragastric balloon combined with diet and exercise (active)
  Interventions: Device: Intragastric balloon device; Procedure: Dietary; Procedure: Exercise intervention

INTERVENTIONS:
Device: Intragastric balloon device — Patients in the experimental arm will benefit from the placement of an Intra Gastric Balloon endoscopically
  Arms: Experimental (BIG + PEC dietary hygiene)
Procedure: Dietary — The patient will benefit from dietary intervention that follows a standard medical recommendation; In consultation with a dietician (at M1, M4, M7, M13, M19, M25), patients will be asked to follow an appropriate diet with a balanced intake of macronutrients (55% carbohydrates, 30% lipids and 15% proteins).
Procedure: Exercise intervention — Patient will benefit from exercise intervention; Resistance and aerobic exercises will be performed twice a week for 3 months (between M4 and M7) under the supervision of a physiotherapist.

SUMMARY:
The aim of this project is to study the effect of an intragastric balloon (IGB) on asthma control in obese patients. Obese patients with uncontrolled asthma will be recruited and randomly assigned to two intervention arms : an intragastric balloon combined with diet and exercise versus diet and exercise alone (control group). The primary endpoint will be the proportion of patients with an improvement based on an Asthma Control Questionnaire (ACQ) score ≥ 0.5 at 1 year compared to baseline.

DETAILED DESCRIPTION:
Asthma and obesity are two major public health problems worldwide. It is now well established that there is a strong link between obesity and asthma. Management of obese patients with asthma is complex in clinical practice because, compared to asthma patients with a normal weight, obese patients with asthma are more prone to respiratory symptoms, asthma attacks and hospital admissions. Lower sensitivity to asthma treatments has also been observed. Indeed, obese patients with moderate to severe asthma respond less well to inhaled corticosteroids, which constitute the recommended treatment for asthma. Improved therapeutic strategies are required for obese patients with uncontrolled asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 65 years
2. Asthma according to the Global Initiative for Asthma (GINA) criteria
3. Patients with uncontrolled asthma based on an ACQ score ≥1.5 despite inhaled corticosteroids ± long acting bronchodilators (LABA)
4. Patients with grade I obesity (BMI> 30 kg/m² and < 35 kg/m²) or morbid obesity (BMI<40 or ≥35 kg/m² with serious physiological risks, as recommended by the French Health Authorities) with contraindications for or refusal of bariatric surgery.
5. Effective contraception for women
6. Patients who have signed a written informed consent form
7. Patients with health insurance
8. Complete COVID-19 vaccination schedule according to current guidelines

Exclusion Criteria:

1. Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
2. Blood eosinophilia greater than 4.5 G/I
3. Treatment by biotherapy within the 12 months after inclusion
4. Cancer diagnosed within the last 5 years
5. Smoking > 10 packs/year (PA)
6. One asthma exacerbation in the 4 weeks leading up to the inclusion visit or IGB placement.
7. Treatment with orlistat Xénical® or GLP1 analogues or regular consumption of narcotics (heroin, cocaine and amphetamines). Analgesic treatments, including level 3, are authorized during the study.
8. Any patient for whom IGB is contraindicated [criteria defined by the French Society for Digestive Endoscopy) and the French Think-Tank for Hepato-Gastroenterology Practices]:

   8.1 Severe cognitive or psychiatric disorders, chronic alcoholism, drug addiction 8.2 Severe and unstabilised eating disorders: bulimia or history of anorexia 8.3 History of gastric surgery including the ring insertion 8.4 Haemostasis disorders 8.5 Anticoagulant or non-steroidal anti-inflammatory medicines 8.6 Severe liver disease 8.7 Pregnancy or desire to become pregnant or breastfeeding 8.8 Anticipated failure to comply with prolonged medical follow-up 8.9 Large hiatal hernias > 5 cm, inflammatory (Crohn's) or stenosing small bowel disease, pyloric stenosis and structural abnormalities of the digestive tract 8.10 Systemic lupus erythematous 8.11 Severe oesophagitis and active gastroduodenal ulcer 8.12 Silicone allergy
9. Patient under guardianship or tutorship, persons placed under the protection of justice or persons participating in another search including an exclusion period still in progress

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Survey | 12 months
  the proportion of patients with changed asthma control at 12 months , defined as a reduction in the Asthma Control Score (ACQ) ≥ 0.5, compared to baseline.

SECONDARY OUTCOMES:
Asthma control | 6 months, 18 months and 24 months
  The proportion of patients with changed asthma control at 6 months, 18 months and 24 months, defined as a reduction in the asthma control score (ACQ) ≥ 0.5 compared to baseline.
Weight loss | 6 months, 12 months, 18 months and 24 months
  Weight loss evaluated according to the percentage weight loss from baseline to post-procedure ([weight before (in kg) - weight after (in kg)] / weight before (in kg)).
The number of patients with an Asthma Control Questionnaire score ≤ 1 | 6 months, 12 months, 18 months and 24 months
  The proportion of patients with an Asthma Control Questionnaire score ≤ 1 measured by ACQ questionnaire
The change of exacerbations | 6 months, 12 months, 18 months and 24 months
  The change of exacerbations which is defined as a course of oral corticosteroids compared to the 12 months period before intervention
The change of hospital admissions or emergency visits for asthma exacerbation | 6 months, 12 months, 18 months and 24 months
  The change in the annual number of hospital admissions or emergency visits for asthma exacerbation compared to baseline with data collection by questionnaire.
Inhaled corticosteroids daily dose | 6 months, 12 months, 18 months, 24 months.
  The change of inhaled corticosteroids daily dose (in ug/d) compared to baseline
Forced expiratory volume in 1 second | 6 months, 12 months, 18 months and 24 months
  The change of forced expiratory volume in 1 second (FEV 1) value measured by plethysmography, and fractions of exhaled nitric oxide (FENO) compared to baseline.
vital capacity | 6 months, 12 months, 18 months and 24 months
  The change of vital capacity value measured by plethysmography, and fractions of exhaled nitric oxide (FENO) compared to baseline.
Total lung capacity | 6 months, 12 months, 18 months and 24 months
  the change of total lung capacity value measured by plethysmography, and fractions of exhaled nitric oxide (FENO) compared to baseline.
Asthma quality | 6 months, 12 months, 18 months and 24 months
  The change of mini-Asthma Quality of Life Questionnaire score compared to baseline.The score is evaluated on 7 points, the highest score indicates a better quality of life

OTHER OUTCOMES:
Physical activity | 6 months, 12 months, 18 months and 24 months
  The change of physical activity score measured by the Ricci and Gagnon Questionnaire compared to baseline. The total score is divided into 3 categories:
  under 18 means inactive physical activity; between 18 and 35 means active physical activity; over 35 means very active activity
Immunoglobulin E (IgE) repertoire of B-lymphocytes | 12 months
  The change of the IgE repertoire of B-lymphocytes compared to baseline: through the gene expression signature profiling of specific IgEs of Der p 1 and Der p 2 (the two main allergens of mites) produced by B cells, using a single cell RNA sequencing technique.

CONTACTS AND LOCATIONS:
Overall Officials: Guilleminault M Laurent, MD, Principal Investigator — Study principal Investigator Toulouse University Hospital
Locations (1):
- University Hospital Toulouse, Toulouse, Occitanie, France